CLINICAL TRIAL: NCT01864187
Title: A Study of the Pharmacokinetics of Dexmedetomidine in Morbid Obesity.
Brief Title: Pharmacokinetics of Dexmedetomidine in Morbid Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Morbid Obesity
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Pharmacokinetics; Dexmedetomidine; Obesity
MeSH Terms: conditions — Obesity | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental): Each team will be administered for 1μg/kg of dexmedetomidine eace one.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The volunteers would receive a dosage of dexmedetomidine by 1μg/kg.

SUMMARY:
Dexmedetomidine hydrochloride ,a relatively new drug in Chinais ,is a highly selective, potent a2-adrenoceptor agonist with significant analgesic, sedative and anxiolytic effects. The morbid obesity in Chinese population is rapidly increasing. But the pharmacokinetics of the drug in these people is still unknown.This research was designed to study the pharmacokinetics of dexmedetomidine in Chinese morbidly obese population.

DETAILED DESCRIPTION:
For the obese are sensitive to the disease such as hypertension, ischaemic heart disease and diabetes, the changes of the state may affect the pharmacokinetics of dexmedetomidine. Besides,the clearance of dexmedetomidine is parallel with liver function and it is excreted by kidney, so differences in the obese may be expected.

About 10 obese patients and 10 matched healthy volunteers with normal weight would be chosen to receive a normal dosage of dexmedetomidine. And venous samples will be collected in different time points. Next the investigators can get the plasma concentration of dexmedetomidine by the use of HPLC-MS. And then the plasma concentration could be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Weight:28≦BMI≦45 and 18.5≦BMI≦24
2. Written informed consent from the patient or the relatives of the participating patient.

Exclusion Criteria:

1. A previous history of intolerance to the study drug or related compounds and additives.
2. Existing significant haematological, endocrine, metabolic or gastrointestinal disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of dexmedetomidine | 0, 5, 10, 15, 20, 25, 30, 45 , 60, 90, 120, 150,180,240,360,480 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Iirola T, Aantaa R, Laitio R, Kentala E, Lahtinen M, Wighton A, Garratt C, Ahtola-Satila T, Olkkola KT. Pharmacokinetics of prolonged infusion of high-dose dexmedetomidine in critically ill patients. Crit Care. 2011;15(5):R257. doi: 10.1186/cc10518. Epub 2011 Oct 26. PMID 22030215
- [Derived] Xu B, Zhou D, Ren L, Shulman S, Zhang X, Xiong M. Pharmacokinetic and pharmacodynamics of intravenous dexmedetomidine in morbidly obese patients undergoing laparoscopic surgery. J Anesth. 2017 Dec;31(6):813-820. doi: 10.1007/s00540-017-2399-y. Epub 2017 Aug 21. PMID 28828532